CLINICAL TRIAL: NCT05309707
Title: ENDOBARC-S Study: "Endovascular Branched Stent-grafts for Aortic ARCh Pathologies in Spain"
Status: Recruiting | Type: Observational
Sponsor: Vascular Investigation Network Spanish Society for Angiology and Vascular Surgery (Network)
Responsible Party: Sponsor
Other Study IDs: 2022-03
Record Dates: First submitted 2022-03-24; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Thoracic Aortic Aneurysm; Thoracic Aortic Dissection; Stent-Graft Endoleak; Stent-Graft Stenosis; Intramural Hematoma; Aortic Diseases; Cardiovascular Diseases; Vascular Diseases
Keywords: Aorta; Thoracic aortic aneurysm; Thoracic aorta dissection; Endovascular repair
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Dissection, Thoracic Aorta; Aortic Diseases; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with aortic arch pathologies treated by branch stent graft systems: Patients with aortic arch pathologies treated by branch stent graft systems (Nexus stent-graft system®, Relay Branch® or Zenith arch branch graft®), with proximal landing at zone 0.
  Interventions: Device: Endovascular exclusion

INTERVENTIONS:
Device: Endovascular exclusion — Endovascular exclusion by branch stent graft systems (Nexus stent-graft system®, Relay Branch® or Zenith arch branch graft®), with proximal landing at zone 0.

SUMMARY:
The ENDOBARC-S post-market clinical follow-up study is undertaken to evaluate the prevention of death related to aortic arch pathologies when treated by branch stent graft systems (Nexus stent-graft system®, Relay Branch® or Zenith arch branch graft®), with proximal landing at zone 0.

The secondary objective is to evaluate the safety and clinical performance of the studied devices.

DETAILED DESCRIPTION:
In this study patients will be observed, who receive a branch stent graft systems (Nexus stent-graft system®, Relay Branch® or Zenith arch branch graft®) for the endovascular treatment of aortic arch pathologies with proximal landing at zone 0. The devices will be implanted at the discretion of the treating physician.

Participating physicians will be asked to provide their observations collected during routine care for patients he/she had decided to treat with the branch stent graft systems for aortic arch (Nexus stent-graft system®, Relay Branch® or Zenith arch branch graft®). Informed consent of the patients to allow the use of their clinical records for the purpose of this observational study will be obtained before data are being collected.

The period of data collection will be approximately 60 months from the index procedure for each patient. Source document verification will be performed on 100% of patients; data from all visits will be reviewed and verified against existing source documents. Complete DICOM image files of the CT scans will be sent to the CoreLab for independent evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 90 years old
* Patient with aortic arch pathologies (aneurysm, pseudoaneurysm, dissection, penetrating ulcer, intramural hematoma), treated by branched stent-grafts (Nexus stent graft system©, Relay® Branch or Zenith arch branch graft®, with proximal landing at zone 0.
* Patient must be available for the appropriate follow-up times for the duration of the study
* Informed consent signed.

Exclusion Criteria:

* Patient less than 18 years old or more than 90 years old.
* Patient has allergies to materials necessary for endovascular repair (e.g. contrast media, anticoagulants or heparin, nitinol, polyester, gold, platinum-iridium)
* Patient has systemic infection or suspected systemic infection
* Patient has thrombocytopenia (platelet count < 150000/µl)
* Patient has untreated hyperthyroidism
* Patient has a progressive or untreated malignancy.
* Patient is pregnant or breastfeeding.
* Patient has a life expectancy of less than 1 year.
* Not informed consent signed

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with aortic arch pathologies (aneurysm, pseudoanerysm, dissection, penetrating ulcer, intramural hematoma), treated by branched stent-grafts (Nexus stent graft system©, Relay® Branch or Zenith arch branch graft®, with proximal landing at zone 0.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Rate of all-cause mortality

SECONDARY OUTCOMES:
Mortality | 24 hours
  Rate of all-cause mortality in peri-operative periods (all related interventions)
Mortality | 3-6, 12, 24, 36, 48, 60 months
  Rate of all-cause mortality
Rupture | 3-6, 12, 24, 36, 48, 60 months
  Rate of patients with aneurysm rupture
Major Adverse Events (MAE) | prior to discharge, 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of patients with major adverse events (aneurysm related death, aneurysm rupture, new myocardial infarction requiring intervention (percutaneous transluminal coronary angioplasty, bypass), new disabling stroke, visceral ischemia (bowel ischemia with surgery or submission to ICU or bowel necrosis with surgery or submission to ICU), new hepatic infarction, new chronic renal insufficiency/renal failure requiring dialysis, new permanent paraplegia, new permanent paraparesis, lower limb ischemia (increase in Rutherford classification) (product-related, procedure-related, aneurysm-related)
Number of interventions | Perioperative
  Rate of interventions in peri-operative periods (all related interventions until index procedure)
Delivery time | Perioperative
  Rate of time intervals the branched-stent graft implantation
Reintervention | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of reinterventions
Endoleak | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of patients with endoleak
Proximal intercomponent separation | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of patients with intercomponent separation at the proximal end of the Nexus stent-graft system > 10 mm
Integrity | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of patients with loss of device integrity (stent fracture and tear in graft material and suture break)
Kinking | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of patients with stent graft or bridging stent graft kinking
Primary patency | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of primary patency of bridging stents
Secondary patency | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of secondary patency of bridging stents
Infection | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of patients with stent graft infection
Primary technical success | 24 hours
  Rate of patients with primary technical success. Technical success is achieved in case all above mentioned criteria are fulfilled, however, an additional unplanned endovascular or surgical procedure is necessitated within 24 h after the index procedure.
  Successful introduction and deployment of the multibranch stent-graft systems in the absence of:
  Surgical conversion Mortality Reintervention Unplanned branch vessel occlusion (post-operative occlusion)
  Including:
  Secure proximal and distal fixation Patent treated branch vessels
Technical success | 24 hours
  Rate of patients with technical success. Technical success is achieved in case all above mentioned criteria are fulfilled, however, an additional unplanned endovascular or surgical procedure is necessitated after the index procedure.
Primary clinical success | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of patients with primary clinical success.
  Primary clinical success is reported on an intent-to-treat basis and is reached if the following criteria are fulfilled at the time of follow-up starting at 12 months follow-up:
  Successful deployment of the endovascular devices at the intended location in the absence of:
  Death as result of aneurysm-related treatment Conversion to open repair Reintervention after index procedure Occlusion of treated branch vessels Type I or III endoleak Increasing aneurysm size Aneurysm rupture
Clinical success | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of patients with clinical success. Clinical success is achieved in case all above mentioned criteria are fulfilled, however, an additional unplanned endovascular or surgical procedure is necessitated after the index procedure.
Stable aneurysm size | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of patients with stable aneurysm size
Decreasing | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of patients with decreasing (<5mm) aneurysm size
Increasing | 30 days, 3-6, 12, 24, 36, 48, 60 months
  Rate of patients with increasing (>5mm) aneurysm size

CONTACTS AND LOCATIONS:
Locations (1):
- Spanish society for Angiology and Vascular Surgery, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Data analyzed by core lab

REFERENCES:
- See also: Spanish Society for Angiology and Vascular Surgery — https://seacv.es